CLINICAL TRIAL: NCT01736540
Title: An Epidemiological Study to Assess the Prevalence of Iron Overload Using MRI in Patients With Transfusional Siderosis (TIMES Study)
Brief Title: An Epidemiological Study to Assess Iron Overload Using MRI in Patients With Transfusional Siderosis (TIMES Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CICL670AAU05
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Results first posted 2016-09-19 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Thalassemia, Non-transfusional-dependent Thalassemia (NTDT), Myeloplastic Dysplasia (MDS), Other Anemia
Keywords: iron overload, liver iron concentration (LIC), cardiac siderosis, transfusional siderosis, magnetic resonance imaging (MRI)
MeSH Terms: conditions — Thalassemia; Iron Overload | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Magnetic Resonance Imaging (MRI) (Other): All participants were subjected to a non-invasive hepatic and cardiac MRI within 60 days of enrollment to measure iron overload.
  Interventions: Device: MRI scan

INTERVENTIONS:
Device: MRI scan — MRI was used to measure both liver and cardiac iron loading (R2 by FerriScan and T2*, respectively).

SUMMARY:
Iron, one of the most common elements in nature and the most abundant transition metal in the body, is readily capable of accepting and donating electrons. This capability makes iron a useful component of various, essential biochemical processes. Despite the essential role of iron, the excess of iron is toxic to the human body. It is critical for the human body to maintain iron balance, since humans have no physiologic mechanism for actively removing iron from the body.

The development of iron overload occurs when iron intake exceeds the body's capacity to safely store the iron in the liver, which is the primary store for iron. Long-term transfusion therapy, a life-giving treatment for patients with intractable chronic anemia is currently the most frequent cause of secondary iron overload.

The mounting evidence regarding the mortality and morbidity due to chronic iron overload in transfusion dependent anaemias has led to the establishment of guidelines that aim the improvement of patient outcomes. Further prospective studies are warranted in order to assess the impact of iron overload in patients with acquired anaemias.

In this study, non-invasive R2- and T2*-MRI techniques were applied to the liver and the heart, respectively, to complement the primary variable (serum ferritin) assessed in patients with various transfusion-dependent anaemias. The main objective of this study was to assess the prevalence and severity of cardiac and liver siderosis in patients with transfusional siderosis. This study was also aim to establish possible correlations between cardiac and liver iron levels with clinical effects in patients with different transfusion-dependent anaemias. Patients were eligible for enrollment irrespective of receiving chelation therapy or not (and irrespective of the chelating agent used).

DETAILED DESCRIPTION:
This study was designed to collect information about a large cohort of patients with anaemias including MDS, aplastic anemia, Diamond-Blackfan, myeloproliferative disorder, as well as haemoglobinopathies (e.g. thalassaemia major, SCD) or other anaemias requiring chronic red blood cell transfusions.

Clinical data was collected retrospectively (if available), unless specified by this protocol (e.g. serum ferritin within less than one month prior to enrollment). All assessments required for this protocol were performed after the patient informed consent is signed. The data was gathered by all study centers and was combined in one central database.

Data was recorded using an electronic case report form (eCRF) at each study site. Adverse events and serious adverse events were recorded for all patients from the date of signed patient informed consent until the MRI tests are performed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Confirmed clinical diagnosis of one of the following disease states: 1. Myelodysplastic syndromes, 2. Thalassaemia major, 3.Other anaemias (e.g. NTDT, SCD, Diamond-Blackfan anaemia, aplastic anaemia, myeloproliferative disease)
* Lifetime history of at least 20 units of red blood cell transfusions AND serum ferritin level > 500 ng/ml; patients with NTDT are not required to have a minimum of 20 units of red blood cell transfusions, but must have serum ferritin level > 300 ng/ml (serum ferritin for all patients must be measured up to 1 month prior to enrollment)
* Written informed consent obtained prior to any procedure required by this protocol

Exclusion Criteria:

Any condition that does not allow the MRI test to be performed: 1. Cardiac pacemaker, 2. Ferromagnetic metal implants other than those approved as safe for use in MR scanners (Example: some types of aneurysm clips, shrapnel), 3. Obesity (exceeding the equipment limits), 4. Patients who are claustrophobic to MR Women who are pregnant Unwillingness or being unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Australia (13):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Wollongong, New South Wales
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, East Bentleigh, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Perth, Western Australia

REFERENCES:
- [Derived] Ho PJ, Hiwase D, Ramakrishna R, Viiala N, Solterbeck A, Traficante R, Zor E, Gervasio OL, High LM, Ross DM, Bowden DK. Cardiac and hepatic siderosis in myelodysplastic syndrome, thalassemia and diverse causes of transfusion-dependent anemia: the TIMES study. Hemasphere. 2019 Jun 4;3(3):e224. doi: 10.1097/HS9.0000000000000224. eCollection 2019 Jun. PMID 31723837

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magnetic Resonance Imaging (MRI)
Started | 243
Completed | 228
Not Completed | 15
Not completed — Did not complete scan within 45 days | 2
Not completed — Death | 1
Not completed — Abnormal test procedure | 1
Not completed — Withdrawal by Subject | 5
Not completed — Protocol Violation | 1
Not completed — Unable to tolerate MRI; claustrophobic | 1
Not completed — No show for MRI appointment | 1
Not completed — Unable to make MRI appointment | 3

BASELINE CHARACTERISTICS:
Arm/Group | Magnetic Resonance Imaging (MRI)
Number analyzed (Participants) | 243
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.8 (20.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 134

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cardiac and Liver Iron Overload.
Description: Hepatic iron overload (liver siderosis) and cardiac iron overload (cardiac siderosis) in patients with transfusional siderosis (Myelodysplastic syndrome (MDS), thalassaemia major, non-transfusion-dependent thalassaemia (NTDT) and other anaemias) were measured using MRI (R2 by FerriScan and T2*, respectively).
Time Frame: 2 months
Population: Only participants with valid T2* by MRI and valid liver iron concentration (LIC) by MRI were included for the cardiac siderosis and liver siderosis analyses, respectively.
Measure: Number; unit: Percentage of participants
Groups:
- Thalassemia Major: Subset of overall participants with thalassemia major
- Melodysplastic Syndrome (MDS): Subset of overall participants with MDS
- Non-transfusion-dependent Anaemia (NTDT): Subset of overall participants with NTDT
- Other Anaemias: Subset of overall participants with other types of anaemia
Arm/Group | Magnetic Resonance Imaging (MRI) | Thalassemia Major | Melodysplastic Syndrome (MDS) | Non-transfusion-dependent Anaemia (NTDT) | Other Anaemias
Number analyzed (Participants) | 228 | 76 | 69 | 18 | 65
Percentage of participants
  Cardiac | 10 | 22 | 4 | 0 | 3
  Liver | 48 | 33 | 55 | 50 | 57

2. Primary Outcome: Cardiac Siderosis Severity
Description: Cardiac siderosis severity was measured by MRI (T2*). The severity grade of siderosis was tiered in 3 levels: mild (T2* >= 20ms), moderate (T2* from 10 to 20ms), and severe (T2* <10ms). Mild cardiac siderosis, by the definitions used in this study, were equivalent to not having cardiac siderosis. Values were compared to published thresholds of iron overload to determine severity of transfusion siderosis in the participant population studied.
Time Frame: 2 months
Population: Only participants with valid T2* by MRI were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Magnetic Resonance Imaging (MRI) | Thalassemia Major | Melodysplastic Syndrome (MDS) | Non-transfusion-dependent Anaemia (NTDT) | Other Anaemias
Number analyzed (Participants) | 228 | 76 | 69 | 18 | 65
Percentage of participants
  None | 89.9 | 77.6 | 95.7 | 100.0 | 95.4
  Moderate | 4.4 | 11.8 | 0.0 | 0.0 | 1.5
  Severe | 5.7 | 10.5 | 4.3 | 0.0 | 3.1

3. Secondary Outcome: Comparison of T2* Levels to Evaluate the Severity of Iron Overload Due to Transfusion Therapy in Chelation-naïve and Chelation-treated Participant Subgroups
Description: Iron overload due to transfusion therapy was assessed based on chelation status of each participant (i.e. minimally exposed to chelator treatment and chelation-treated patient subgroups).
Time Frame: 2 months
Population: Only participants with valid T2* by MRI were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: ms
Arm/Group | Magnetic Resonance Imaging (MRI) | Thalassemia Major | Melodysplastic Syndrome (MDS) | Non-transfusion-dependent Anaemia (NTDT) | Other Anaemias
Number analyzed (Participants) | 228 | 76 | 69 | 18 | 65
ms
  Overall (n=228,76,69,18,65) | 30.2 [27.62 to 32.62] | 23.95 [21.46 to 26.72] | 30.13 [26.78 to 33.90] | 32.69 [25.94 to 41.19] | 30.76 [27.29 to 34.67]
  Chelation naïve/minimally exposed(n=75,0,27,11,37) | 32.55 [28.71 to 36.91] | NA [NA to NA] — No participants were minimally exposed to chelator treatment. | 32.05 [26.66 to 38.53] | 32.95 [24.70 to 43.97] | 32.66 [27.91 to 38.22]
  Chelator exposed (n=153,76,42,7,28) | 28.25 [25.28 to 31.57] | 23.95 [21.46 to 26.72] | 28.32 [24.43 to 32.82] | 32.43 [22.59 to 46.55] | 28.96 [24.17 to 34.70]

4. Secondary Outcome: Comparison of Liver Iron Concentration (LIC) Levels to Evaluate Iron Overload Due to Transfusion Therapy in Chelation-naïve and Chelation-treated Participant Subgroups
Description: Iron overload due to transfusion therapy was assessed based on chelation status of each participant (i.e. minimally exposed to chelator treatment and chelation-treated patient subgroups). The mean data presented are mean estimates of log transformed data.
Time Frame: 2 months
Population: Only participants with valid LIC by MRI were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: mg Fe/g
Arm/Group | Magnetic Resonance Imaging (MRI) | Thalassemia Major | Melodysplastic Syndrome (MDS) | Non-transfusion-dependent Anaemia (NTDT) | Other Anaemias
Number analyzed (Participants) | 228 | 76 | 69 | 18 | 65
mg Fe/g
  Overall (n=228,76,69,18,65) | 11.30 [9.42 to 13.17] | 8.09 [5.62 to 10.57] | 10.84 [8.18 to 13.50] | 12.38 [7.16 to 17.59] | 12.28 [9.58 to 14.98]
  Chelation naïve/minimally exposed(n=75,0,27,11,37) | 8.73 [5.90 to 11.56] | NA [NA to NA] — No participants were minimally exposed. | 10.28 [6.13 to 14.43] | 5.00 [-1.50 to 11.50] | 10.92 [7.37 to 14.47]
  Chelator exposed (n=153,76,42,7,28) | 13.22 [10.72 to 15.72] | 8.09 [5.62 to 10.57] | 11.40 [8.07 to 14.72] | 19.76 [11.60 to 27.91] | 13.64 [9.56 to 17.72]

5. Secondary Outcome: Mean Serum Ferritin According to the Presence or Absence of Retrospective Cardiac Events
Description: Mean serum ferritin according to the presence or absence of cardiac events was assessed for all participant subgroups.
Time Frame: 12 months - retrospective
Population: Participants with serum ferritin values and previous cardiac events data were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Magnetic Resonance Imaging (MRI)
Number analyzed (Participants) | 238
ng/mL
  Cardiac event in past 12 months = yes (n=12) | 2153.6 (1878.6)
  Cardiac event in past 12 months = no (n=226) | 2150.2 (1914.5)

6. Secondary Outcome: Mean Serum Ferritin According to the Presence or Absence of Retrospective Hepatic Events
Description: Mean serum ferritin according to the presence or absence of hepatic events was assessed for all participant subgroups.
Time Frame: 12 months - retrospective
Population: Participants with serum ferritin values and previous hepatic events data were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Magnetic Resonance Imaging (MRI)
Number analyzed (Participants) | 239
ng/mL
  Hepatic event in the past 12 months = yes (n=8) | 3302.8 (2684.3)
  Hepatic event in the past 12 months = no (n=231) | 2124.1 (1879.2)

7. Secondary Outcome: Mean Cardiac T2* According to the Presence or Absence of Retrospective Cardiac Events
Description: Mean cardiac T2* according to the presence or absence of cardiac events was assessed for all participant subgroups. The mean data presented are mean estimates of log transformed data.
Time Frame: 12 months - retrospective
Population: Participants with valid T2* by MRI results were included in the analysis.
Measure: Mean (Standard Deviation); unit: log10 (ms)
Arm/Group | Magnetic Resonance Imaging (MRI)
Number analyzed (Participants) | 228
log10 (ms)
  Cardiac event in past 12 months = yes (n=12) | 1.546 (0.0979)
  Cardiac event in the past 12 months = no (n=226) | 1.445 (0.2188)

8. Secondary Outcome: Mean LIC According to the Presence or Absence of Retrospective Hepatic Events
Description: Mean LIC according to the presence or absence of hepatic events was assessed for all participant subgroups.
Time Frame: 12 months - retrospective
Population: Participants with LIC by MRI were included in the analysis.
Measure: Mean (Standard Deviation); unit: mg Fe/g
Arm/Group | Magnetic Resonance Imaging (MRI)
Number analyzed (Participants) | 228
mg Fe/g
  Hepatic event in past 12 months = yes (n=7) | 17.51 (15.292)
  Hepatic event in past 12 months = no (n=221) | 10.08 (10.950)

9. Secondary Outcome: Mean Blood Magnetic Susceptibility (BMS)
Description: Blood samples were collected to assess BMS. The measurement represents absolute magnetic susceptibility at 1 month. Whole blood magnetic susceptibility was calculated by the addition of the dry weight susceptibility and the contribution of the water driven from the sample.
Time Frame: 1 month
Population: Participants with BMS values were analyzed.
Measure: Mean (Standard Deviation); unit: emu/g wet wt/Oe
Arm/Group | Magnetic Resonance Imaging (MRI)
Number analyzed (Participants) | 233
emu/g wet wt/Oe | -6.18 (0.147)

10. Secondary Outcome: Percentage of Participants Transfused With Erythrocytes
Description: Transfusion requirement in participants with acquired anaemias with history of receiving chelation therapy was assessed.
Time Frame: 12 months - retrospective
Population: Participants with a erythrocyte transfusion history were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Magnetic Resonance Imaging (MRI) | Thalassemia Major | Melodysplastic Syndrome (MDS) | Non-transfusion-dependent Anaemia (NTDT) | Other Anaemias
Number analyzed (Participants) | 241 | 81 | 73 | 19 | 68
Percentage of participants | 95.0 | 100.0 | 100.0 | 36.8 | 100.0

11. Secondary Outcome: Percentage of Participants With Time Since Most Recent Transfuison of <7 Days, 7 to < 14 Days, 14 to < 30 Days, 30 to < 60 Days or >= 60 Days
Description: Transfusion requirement in participants with acquired anaemias with history of receiving chelation therapy was assessed.
Time Frame: 12 months - retrospective
Population: Participants with data on time since their most recent transfusion were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Magnetic Resonance Imaging (MRI) | Thalassemia Major | Melodysplastic Syndrome (MDS) | Non-transfusion-dependent Anaemia (NTDT) | Other Anaemias
Number analyzed (Participants) | 241 | 81 | 68 | 19 | 65
percentage of participants
  < 7 days | 43.1 | 72.8 | 31.0 | 14.3 | 22.7
  7 - < 14 days | 12.9 | 2.5 | 28.2 | 14.3 | 9.1
  14 - < 30 days | 20.0 | 22.2 | 14.1 | 0.0 | 25.8
  30 - < 60 days | 5.8 | 2.5 | 9.9 | 14.3 | 4.5
  >= 60 days | 18.2 | 0.0 | 16.9 | 57.1 | 37.9

12. Secondary Outcome: Mean Number of Erythrocyte Units Transfused in Last 12 Months
Description: Transfusion requirement in participants with acquired anaemias with history of receiving chelation therapy was assessed.
Time Frame: 12 months - retrospective
Population: Participants with 'number of units transfused' data were included in the analysis.
Measure: Mean (Standard Deviation); unit: number of units transfused
Arm/Group | Magnetic Resonance Imaging (MRI) | Thalassemia Major | Melodysplastic Syndrome (MDS) | Non-transfusion-dependent Anaemia (NTDT) | Other Anaemias
Number analyzed (Participants) | 228 | 81 | 72 | 7 | 68
number of units transfused | 33.3 (21.0) | 41.4 (9.5) | 34.7 (25.6) | 8.4 (12.2) | 24.8 (21.5)

13. Secondary Outcome: Mean Quality of Life (QOL) Scores
Description: Quality of life was assessed using the Short Form 36 (SF-36) Health Survey. The SF-36 consists of 8 sub-scales: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. The raw sores of the 8 scales are transformed to a 0 - 100 scale where 0 indicates maximum disability and 100 indicates no disability. There also are two physical and mental health summary measures. Each summary measure is the mean average of the 4 associated sub-scale scores. The range for each summary measure is 0 to 100 where 0 represents maximum disability and 100 represents no disability.
Time Frame: 1 month
Population: Only participants with data for each subscale were included in the analysis for that subscale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Magnetic Resonance Imaging (MRI) | Thalassemia Major | Melodysplastic Syndrome (MDS) | Non-transfusion-dependent Anaemia (NTDT) | Other Anaemias
Number analyzed (Participants) | 243 | 81 | 74 | 20 | 68
units on a scale
  Physical functioning | 43.10 (11.471) | 49.79 (9.144) | 35.67 (9.791) | 49.37 (7.576) | 41.56 (11.139)
  Role physical | 42.54 (10.895) | 49.51 (8.836) | 36.71 (9.462) | 46.46 (8.717) | 39.44 (10.229)
  Bodily pain | 48.41 (10.969) | 50.48 (11.084) | 45.52 (10.750) | 54.66 (7.773) | 47.60 (10.815)
  General health | 41.65 (9.909) | 44.82 (9.365) | 39.48 (9.595) | 43.23 (8.893) | 39.80 (10.239)
  Vitality | 45.59 (10.267) | 50.18 (9.277) | 42.41 (9.190) | 48.95 (8.424) | 42.67 (10.757)
  Social functioning | 44.99 (11.075) | 48.98 (9.869) | 42.37 (10.486) | 46.43 (9.905) | 42.67 (12.043)
  Role emotional | 43.83 (12.977) | 48.99 (11.236) | 40.11 (13.101) | 47.03 (10.552) | 40.89 (13.320)
  Mental health | 47.84 (11.149) | 50.09 (11.240) | 46.69 (9.495) | 48.74 (9.846) | 46.12 (12.632)
  Physical component summary | 43.48 (9.808) | 48.75 (7.809) | 37.55 (8.748) | 50.34 (6.392) | 41.93 (9.524)
  Mental component summary | 46.76 (11.622) | 49.58 (10.354) | 45.91 (10.349) | 47.47 (10.832) | 44.08 (13.822)

14. Secondary Outcome: Percentage of Participants With Low Medium or High Adherence to Iron Chelator Therapy
Description: Adherence of participants was assessed using an adherence questionnaire. Adherence questionnaires were completed only by participants who received chelating agents. Participants answered yes or no to 6 statements such as "Forgot to take pills". Based on the responses to these questions, adherence was classified as low, medium or high.
Time Frame: 1 month
Population: Participants who were on iron chelator therapy at screening, and had answered at least one question on the questionnaire and had sufficient information to score the questionnaire, were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Magnetic Resonance Imaging (MRI) | Thalassemia Major | Melodysplastic Syndrome (MDS) | Non-transfusion-dependent Anaemia (NTDT) | Other Anaemias
Number analyzed (Participants) | 141 | 78 | 34 | 4 | 25
Percentage of participants
  Low | 27.7 | 32.1 | 11.8 | 75.0 | 28.0
  Medium | 61.7 | 57.7 | 73.5 | 25.0 | 64.0
  High | 10.6 | 10.3 | 14.7 | 0.0 | 8.0

15. Secondary Outcome: Investigator Treatment Decisions Based on MRI Results
Description: Treatment decisions were recorded after the investigator evaluated the MRI results, in order to assess the impact of such diagnostic test on the overall clinical management of participants with iron overload. Investigators answered the following question: "Since the MRI scan, have you changed or are planning to change the management of iron in your subject?".
Time Frame: 2 months
Population: Participants, for whom treatment decision questionnaire results were provided and for whom MRI results were available, were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Magnetic Resonance Imaging (MRI)
Number analyzed (Participants) | 229
Percentage of participants
  Answer = yes | 42.4
  Answer = no | 57.6

ADVERSE EVENTS:
Groups:
- Thalassaemia Major: Subset of overall participants with thalassemia major
- Myelodysplastic Syndrome (MDS): Subset of overall participants with MDS
- Other Anaemia: Subset of overall participants with other types of anaemias
Arm/Group | Thalassaemia Major | Myelodysplastic Syndrome (MDS) | Other Anaemia | Non-transfusion-dependent Anaemia (NTDT)
Serious Adverse Events (participants affected / at risk) | 2/81 | 8/74 | 2/68 | 0/20
Other Adverse Events (participants affected / at risk) | 7/81 | 9/74 | 3/68 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thalassaemia Major (N=81) | Myelodysplastic Syndrome (MDS) (N=74) | Other Anaemia (N=68) | Non-transfusion-dependent Anaemia (NTDT) (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Medical device site erosion (General disorders) | 1 | 0 | 0 | 0
Medical device site pain (General disorders) | 1 | 0 | 0 | 0
Medical device site swelling (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thalassaemia Major (N=81) | Myelodysplastic Syndrome (MDS) (N=74) | Other Anaemia (N=68) | Non-transfusion-dependent Anaemia (NTDT) (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.